CLINICAL TRIAL: NCT02738801
Title: Randomized, Double-Blind, Parallel Group, Placebo-Controlled, Multicenter, Exploratory Phase IIa Study to Assess Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of GLPG1690 Administered for 12 Weeks in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Study to Assess Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of GLPG1690 in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1690-CL-202; 2015-004157-41 (EudraCT Number)
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; GLPG1690; Autotaxin
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — GLPG1690

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG1690 600 mg once daily (QD) (Experimental)
  Interventions: Drug: GLPG1690 600 mg QD
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo QD

INTERVENTIONS:
Drug: GLPG1690 600 mg QD — GLPG1690 capsules, administered at a dose of 600 mg, orally QD
  Arms: GLPG1690 600 mg once daily (QD)
Drug: Placebo QD — Matching placebo capsules, administered orally QD
  Arms: Placebo QD

SUMMARY:
A multicenter randomized, double-blind, parallel group, placebo-controlled, exploratory phase IIa study in subjects with Idiopathic Pulmonary Fibrosis (IPF) to evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of GLPG1690. Male and female subjects aged 40 years or older will be screened to determine eligibility. The screening period will be up to 4 weeks. At baseline, eligible subjects will be randomized in a 3:1 ratio to GLPG1690 or matching placebo administered for 12 weeks. The subjects will visit the study center at screening, baseline, Weeks 1, 2, 4, 8 and 12 and for a follow-up visit 2 weeks after the last administration of study drug. Planned assessments: Adverse event reporting, clinical laboratory tests, vital signs, physical examination, 12-Lead-ECG, PK blood sampling, biomarker blood/bronchoalveolar lavage fluid (BALF), Spirometry, St George's respiratory questionnaire, high-resolution computed tomography (HRCT).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able and willing to sign the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved Informed Consent Form (ICF)
2. Male or female subjects of non-child-bearing potential aged ≥ 40 years
3. Subjects with a chest HRCT performed within 12 months prior to screening
4. Subjects with IPF diagnosed by a multidisciplinary team
5. Subjects with: a. forced vital capacity (FVC) ≥50% predicted of normal AND b. Diffusing capacity for the lungs for carbon monoxide (DLCO) ≥ 30% predicted of normal corrected for hemoglobin
6. Subjects with a forced expiratory volume in 1 second (FEV1)/FVC (Tiffeneau-Pinelli index) ratio ≥ 0.70 (based on pre-bronchodilator spirometry
7. Subjects on stable supportive care
8. Subjects in stable condition

Exclusion Criteria:

1. Subjects with know hypersensitivity to any of the study drug ingredients
2. Subjects with a history of or current immunosuppressive condition
3. Subjects with a history of malignancy within the past 5 years
4. Subjects with clinically significant abnormalities on ECG
5. Subjects with acute IPF exacerbation within 6 weeks prior to screening
6. Subjects with a lower respiratory tract infection requiring antibiotics with 4 weeks prior to screening
7. Smoking within 3 months pre-screening
8. Interstitial lung disease
9. History of lung volume reduction surgery or lung transplant
10. Unstable cardiac or pulmonary disease other than IPF within 6 months prior to screening
11. Subjects with abnormal liver function
12. Subjects with abnormal renal function

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Fieuw, MD, Study Director — Galapagos NV
Locations (8):
- Ukraine (6):
  - Municipal Clinical Hospital # 6, Dnipropetrovsk
  - Kharkov City Clinical Hospital # 13, Kharkiv
  - F.G. Yanovskyy Institute of Phthisiatry and Pulmonology 1, Kiev
  - F.G. Yanovskyy Institute of Phthisiatry and Pulmonology 2, Kiev
  - Oesa Regional Clinical Hospital, Odesa
  - Poltava Regional Clinical Antituberculosis Dispancery, Poltava
- United Kingdom (2):
  - Royal Brompton Hospital, London
  - The Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maher TM, van der Aar EM, Van de Steen O, Allamassey L, Desrivot J, Dupont S, Fagard L, Ford P, Fieuw A, Wuyts W. Safety, tolerability, pharmacokinetics, and pharmacodynamics of GLPG1690, a novel autotaxin inhibitor, to treat idiopathic pulmonary fibrosis (FLORA): a phase 2a randomised placebo-controlled trial. Lancet Respir Med. 2018 Aug;6(8):627-635. doi: 10.1016/S2213-2600(18)30181-4. Epub 2018 May 20. PMID 29792287

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Once Daily (QD): Participants received matching oral capsules QD for 12 weeks.
- GLPG1690 600 mg QD: Participants received 600 mg GLPG1690, administered as oral capsules QD for 12 weeks.
Period: Overall Study
Arm/Group | Placebo Once Daily (QD) | GLPG1690 600 mg QD
Started | 6 | 17
Completed | 5 | 15
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all randomized participants who received at least one dose of GLPG1690.
Groups:
- Placebo QD: Participants received matching oral capsules QD for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo QD | GLPG1690 600 mg QD | Total
Number analyzed (Participants) | 6 | 17 | 23
Age, Continuous [Median (Full Range); unit: years] | 64.0 [52 to 72] | 67.0 [54 to 79] | 66.0 [52 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 17 | 23
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-Emergent Adverse Events (AEs)
Time Frame: From screening up to Day 98
Population: Safety Population: all randomized participants who received at least one dose of GLPG1690.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD | GLPG1690 600 mg QD
Number analyzed (Participants) | 6 | 17
Participants | 4 | 11

2. Primary Outcome: Mean Maximum Observed Plasma Concentration (Cmax; Micrograms Per Milliliter [µg/mL]) of GLPG1690
Time Frame: Baseline, predose on Days 7, 14, 28, 56, 84, and 98 (or at early discontinuation), and at 1.5, 4, and 6 hours postdose on Day 28
Population: Pharmacokinetic (PK) Analysis Set: all randomized participants who received at least one dose of GLPG1690 and for whom evaluable PK data were available. Excludes 1 patient who withdrew because of an AE prior to Week 1 (and had only PK concentrations for baseline and early discontinuation) and 1 patient with only a single predose sample at Week 4
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | GLPG1690 600 mg QD
Number analyzed (Participants) | 15
µg/mL | 6.06 (4.92)

3. Primary Outcome: Median Time to Occurrence of GLPG1690 Cmax (Tmax; Hours [h])
Time Frame: as for outcome 2
Population: PK Analysis Population; excludes 1 patient who withdrew because of an AE prior to Week 1 (and had only PK concentrations for baseline and early discontinuation) and 1 patient with only a single predose sample at Week 4.
Measure: Median (Full Range); unit: hours
Arm/Group | GLPG1690 600 mg QD
Number analyzed (Participants) | 15
hours | 4 [1.5 to 6]

4. Primary Outcome: Mean Area Under the Plasma Concentration-Time Curve (AUC[t]; µg.h/mL) of GLPG1690
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg.h/mL
Arm/Group | GLPG1690 600 mg QD
Number analyzed (Participants) | 15
µg.h/mL | 55.6 (46.6)

5. Primary Outcome: Mean GLPG1690 Plasma Concentration Observed at Predose (Ctrough; µg/mL)
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | GLPG1690 600 mg QD
Number analyzed (Participants) | 15
µg/mL | 0.624 (0.846)

6. Primary Outcome: Mean Peak Area Ratio of Lysophosphatidic Acid (LPA) C18:2 Species in Blood
Description: LPA species C18:2 concentrations were determined in blood using a validated liquid chromatography tandem mass spectometry (LC/MS-MS) method. The baseline reference timepoint was Day -1 (mean of the pre-dosing duplicates).
Time Frame: Baseline (Day -1), predose and 1.5 and 6 hours postdose on Day 28, predose on Day 84, and Day 98 (or early discontinuation)
Population: Pharmacodynamic (PD) Population: all randomized participants who received at least one dose of GLPG1690 and had at least one postbaseline assessment with PD data. Only patients with assessments at both baseline and the pre-specified visit(s) were included in the analysis.
Measure: Mean (Standard Error); unit: peak area ratio
Arm/Group | Placebo QD | GLPG1690 600 mg QD
Number analyzed (Participants) | 6 | 17
peak area ratio
  Baseline | 0.4180 (0.1088) | 0.3311 (0.0670)
  Day 28: number analyzed (Participants) | 5 | 16
  Day 28 | 0.3650 (0.0895) | 0.1476 (0.0380)
  Day 28 (1.5 hours postdose): number analyzed (Participants) | 5 | 15
  Day 28 (1.5 hours postdose) | 0.4071 (0.1352) | 0.0479 (0.0120)
  Day 28 (6 hours postodse): number analyzed (Participants) | 5 | 15
  Day 28 (6 hours postodse) | 0.3402 (0.1373) | 0.0314 (0.0046)
  Day 84: number analyzed (Participants) | 6 | 15
  Day 84 | 0.4080 (0.1090) | 0.0898 (0.0160)
  Day 98: number analyzed (Participants) | 5 | 15
  Day 98 | 0.4672 (0.1647) | 0.5172 (0.1660)

7. Primary Outcome: Mean Peak Area Ratio of LPA C18:2 Species in Bronchoalveolar Lavage Fluid (BALF)
Description: LPA species C18:2 concentrations were determined in BALF using a validated LC/MS-MS method. The baseline reference timepoint was Day -1 (mean of the pre-dosing duplicates).
Time Frame: Baseline (Day -1) and Day 84
Population: PD Population; only patients with assessments at both baseline and the pre-specified visit were included in the analysis.
Measure: Mean (Standard Error); unit: peak area ratio
Arm/Group | Placebo QD | GLPG1690 600 mg QD
Number analyzed (Participants) | 6 | 17
peak area ratio
  Baseline | 0.0026 (0.0011) | 0.0009 (0.0002)
  Day 84: number analyzed (Participants) | 5 | 14
  Day 84 | 0.0035 (0.0028) | 0.0011 (0.0002)

ADVERSE EVENTS:
Time Frame: From Screening to final follow-up visit (Day 98)
Arm/Group | Placebo QD | GLPG1690 600 mg QD
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/17
Other Adverse Events (participants affected / at risk) | 4/6 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=6) | GLPG1690 600 mg QD (N=17)
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=6) | GLPG1690 600 mg QD (N=17)
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2
Infected cyst (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Electrocardiogram PR prolongation (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must agree that before publishing or communicating any results of the trial, the sponsor has at least 60 days for full review of the information prior to submission.

DOCUMENTS (2):
  • Study Protocol (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT02738801/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT02738801/SAP_001.pdf